CLINICAL TRIAL: NCT03895424
Title: An Iron Isotope Study in Humans to Evaluate the Iron Bioavailability of a Novel Iron Compound - Iron Fatty Acid Complex
Brief Title: Iron Isotope Study of an Iron Fatty Acid Complex
Acronym: IFAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IFAC
Record Dates: First submitted 2019-03-07; First posted 2019-03-29 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Iron-deficiency
Keywords: Iron; Isotope study; Fatty Acid
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron Fatty Acid Complex (IFAC) (Experimental): The iron fatty acid complex encapsulated and administered to the participants
  Interventions: Dietary Supplement: IFAC
- Micellarized iron fatty acid complex (MIFAC) (Experimental): Micellarized form of the iron fatty acid complex which is enscapsulated and administered to the participants
  Interventions: Dietary Supplement: MIFAC
- Control Ferrous Sulfate (Active Comparator): Ferrous sulfate that is provided in the form of a solution along with a capsule that contains the same amount of fat that is present in the other two arms.
  Interventions: Dietary Supplement: Control Ferrous Sulfate

INTERVENTIONS:
Dietary Supplement: IFAC — This intervention will contain the iron fatty acid complex in a capsule. The complex will be labelled with the iron isotope 58Fe
  Arms: Iron Fatty Acid Complex (IFAC)
Dietary Supplement: MIFAC — This intervention will contain the micellarized form of the iron fatty acid complex in a capsule. The complex will be labelled with the iron isotope with 57Fe
  Arms: Micellarized iron fatty acid complex (MIFAC)
Dietary Supplement: Control Ferrous Sulfate — This intervention will contain ferrous sulfate in the form of a solution labelled with the iron isotope 54Fe. A capsule with the same amount of fat as in the other arms will be administered to the participants
  Arms: Control Ferrous Sulfate

SUMMARY:
The study aims at assessing the iron (Fe) bioavailability from a newly developed iron compound - an iron fatty acid complex. The iron from the compound is hypothesized to have a higher absorption rate than commonly available supplements in the market. The study is a cross over, human iron isotope study with three arms where participants consume the experimental dietary products in a randomized fashion. The study duration is of 45 days - from the day of the capsule administration till the last blood sampling point

DETAILED DESCRIPTION:
Iron deficiency remains a major public health concern in both industrialized and non-industrialized (developing) countries. Most supplements in the present day, to address the problem of iron deficiency, are in the form of ferrous salts, especially ferrous sulfate. Ferrous salts are absorbed by the non-heme iron pathway involving the Divalent Metal Transporter 1 (DMT-1) receptor, where the absorption rate is 20% of the total iron content. The common strategy of the food supplement industries is to increase the iron load in the supplements to provide the necessary amount of iron, compensating for the low absorption rate. However, these have side effects associated with the high dosage. Instead of a high dosage, a more effective strategy would be to incorporate the iron in a way that the absorption rate is maximized. The intervention product, an iron fatty acid complex (IFAC), containing 12 mg of iron, is expected to be absorbed as effective as any ferrous sulfate supplement in the market due to the alternative metabolic route that is hypothesized to be taken by the complex.

The first week of the study comprises of the administration of the capsules containing the complexes to the participants on day 1 , day 3 and day 5 of the study respectively. Blood samples are collected on day 10,20, 30 and 40 and 160 days after the last day of the capsule administration..

The primary objectives of this trial are:

To assess the iron bioavailability from the developed iron salt fatty acid complexes (IFAC) and micro-emulsified iron fatty acid complex (MIFAC) and compare it with the bioavailability of the reference ferrous sulfate (FeSO4) To investigate whether the MIFAC promotes absorption compared to IFAC and the reference.

Fractional iron absorption from the three intervention products will be calculated based on the shift of the stable iron isotope ratios in collected blood samples at 10, 20, 30, 40 and 160 days after administration of the stable isotopically labelled capsules. Stable iron isotope ratios will be determined by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 - 40 years old
* marginal iron status (ferritin <25 ng/ml; measured by study coordinator)
* body weight up to 65 kg
* normal body mass index (bodyweight [kg] / (height [m])2 = 18.5 - 25)
* do not take any vitamin or mineral supplements two weeks before and during the study.
* do not have a metabolic, gastrointestinal or chronic diseases
* able to communicate in and comprehend English language

Exclusion Criteria:

* pregnant or breast-feeding
* on long-term medication (except oral contraceptive)
* elevated C-reactive Protein (>5mg/L; will be measured by study coordinator)
* medium or strong anemic (hemoglobin <9.0 g/dL; will be measured by study coordinator)
* donated blood within the last 4 months before the study start date
* taking part in another clinical study at the same time or had within the last 30 days before the study date
* participated in an earlier study using iron stable isotopes.
* eating disorder or a strong allergy.
* cannot be expected to comply with study protocol (e.g. not available on certain study appointments or difficulties with blood sampling)
* unable to understand the information sheet and the informed consent form due to cognitive or language reasons

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females are allowed to participate in the study
Enrollment: 29 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption from IFAC | Day 10 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from IFAC | Day 20 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from IFAC | Day 30 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from IFAC | Day 40 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from IFAC | Day 160 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from MIFAC | Day 10 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from MIFAC | Day 20 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from MIFAC | Day 30 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from MIFAC | Day 40 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from MIFAC | Day 160 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from Control Ferrous Sulfate | Day 10 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from Control Ferrous Sulfate | Day 20 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from Control Ferrous Sulfate | Day 30 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from Control Ferrous Sulfate | Day 40 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.
Fractional iron absorption from Control Ferrous Sulfate | Day 160 of the study
  The primary outcome is the fractional iron absorption, which will be compared in predefined comparisons from the three different capsules that will be administered to the study participants. Relative bioavailability, defined as the ratio of fractional absorption relative to the reference dose (absorption measured from encapsulated FeSO4), will be also compared in predefined comparisons.

SECONDARY OUTCOMES:
Haemoglobin | Day 1 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Haemoglobin | Day 10 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Haemoglobin | Day 20 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Haemoglobin | Day 30 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Haemoglobin | Day 40 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Haemoglobin | Day 160 of the study
  Haemoglobin status of the participants will be measured to check for anaemia status
Ferritin | Day 1 of the study
  Ferritin levels will be measured to assess the iron stores in the participants.
Ferritin | Day 10 of the study
  Ferritin levels will be measured to assess the iron stores in the participants.
Ferritin | Day 20 of the study
  Ferritin levels will be measured to assess the iron stores in the participants.
Ferritin | Day 30 of the study
  Ferritin levels will be measured to assess the iron stores in the participants.
Ferritin | Day 40 of the study
  Ferritin levels will be measured to assess the iron stores in the participants.
C-reactive Protein | Day 1 of the study
  Inflammation status of the participants will be measured since it has an effect on iron absorption
C-reactive Protein | Day 10 of the study
  Inflammation status of the participants will be measured since it has an effect on iron absorption
C-reactive Protein | Day 20 of the study
  Inflammation status of the participants will be measured since it has an effect on iron absorption
C-reactive Protein | Day 30 of the study
  Inflammation status of the participants will be measured since it has an effect on iron absorption
C-reactive Protein | Day 40 of the study
  Inflammation status of the participants will be measured since it has an effect on iron absorption

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, PhD, Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- Lab of Human Nutrition, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided